CLINICAL TRIAL: NCT01733212
Title: Efficacy of Ginger on Intraoperative and Postoperative Nausea and Vomiting in Elective Cesarean Section Patients.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Joel Yarmush (Other)
Responsible Party: Sponsor-Investigator, Joel Yarmush, Attending Physician, Program Director (Anesthesiology), New York Presbyterian Brooklyn Methodist Hospital
Organization: New York Presbyterian Brooklyn Methodist Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB:147810
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Results first posted 2018-05-11 (Actual); Last update posted 2021-09-10 (Actual); Status verified 2018-08

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting; Cesaraen; Ginger; cesarean section
MeSH Terms: conditions — Nausea; Vomiting | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger (Experimental): 2 gm powder of ginger filled in a capsule
  Interventions: Drug: Ginger
- Placebo (Placebo Comparator): 2 gm of placebo pill (A capsule)
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Ginger — Ginger is an herb. The rhizome (underground stem) is used as a spice and also as a medicine. It can be used fresh, dried and powdered, or as a juice or oil. Two capsules (1g each) of dry powdered ginger are given, one capsule a half-hour before induction of anesthesia and the second 2h after surgery.
  Other Names: Zingiber Officinale
  Arms: Ginger
Drug: Placebo Oral Tablet — Two capsules (1g each) of placebo, one capsule a half-hour before induction of anesthesia and the second 2h after surgery.
  Arms: Placebo

SUMMARY:
SPECIFIC AIMS

* Assess risk factors for nausea and vomiting in c-section patients undergoing regional anesthesia
* Quantify the incidence of nausea and vomiting intraoperatively and postoperatively in the ginger and placebo groups.
* Quantify post-operative analgesia and pruritus in the ginger and placebo groups
* Quantify patient satisfaction of the ginger and placebo groups
* Assess patient expectation of ginger on post-op day three

DETAILED DESCRIPTION:
Two hundred and thirty nine ASA class I and II patients, scheduled for elective c-section will be assigned randomly to receive either 1g ginger tablet PO (Group 1) or 1 g placebo PO (Group 2) preoperatively, immediately before surgery. The usual preoperative anti-emetic and antacid regimen will be continued for both groups. Initial blood pressure, pulse and hemoglobin and hematocrit will be documented by the researcher prior to the arrival of the patient into the operating room. A baseline questionnaire will be given to the patients to assess risk factors for nausea and vomiting. Questions will include: age, BMI, parity, weeks gestation, h/o seasickness, h/o of hyperemesis gravidrum in this or prior pregnancies, h/o PONV, medical problems, any medication used within past 24 hrs, education and occupation.

Intraoperatively, both groups will receive combined spinal-epidural anesthesia in the usual manner. All standard monitoring will be applied and vital signs recorded for the entirety of the procedure. The number and dose of ephedrine or phenylephrine boluses and the number and severity of nausea episodes (using a Visual Analog Scale (VANS)) and number of vomiting episodes will be noted. In addition the following will be recorded: if uterus was exteriorized, any medications used by the anesthesiologist (other than ephedrine and phenylephrine), and estimated blood loss.

Postoperatively, patients will receive either a one time dose of the 1g ginger PO (Group 1) or 1 g placebo PO (Group 2) 2 hours after entering the postanesthesia care unit (PACU). Thirty minutes after the medication is given, patients will be asked to rate their nausea, level of analgesia, and level of pruritus on a VANS, and vomiting episodes will be recorded. Medications given for nausea will be continued in the post-operative period for both groups. The doses of Zofran will be counted in the 24 hr postoperative period. Twenty-four hours after surgery, blood will be drawn to assess hemoglobin and hematocrit as well as to assess platelet function.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (i.e., ASA I, or II) patients presenting for planned c-section at New York Methodist Hospital
* Signed informed consent

Exclusion Criteria:

* They are unable or unwilling to take part in the study
* They have a history of an allergy to any medications used including ginger
* They have had any gastrointestinal surgery on the stomach, small intestine, or gall bladder.
* They have any history of bleeding disorder, (i.e., Hemophilia A/B, ITP, etc.)
* They have a contraindication to intrathecal or epidural anesthesia. ( i.e., Arnold- Chiari malformation, etc.)
* They are unable to understand instructions or questions related to study
* ASA III or IV patients

Ages: 20 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Weinberg, MD, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Methodist Hospital, Brooklyn, New York, United States

REFERENCES:
- [Derived] Griffiths JD, Gyte GM, Popham PA, Williams K, Paranjothy S, Broughton HK, Brown HC, Thomas J. Interventions for preventing nausea and vomiting in women undergoing regional anaesthesia for caesarean section. Cochrane Database Syst Rev. 2021 May 18;5(5):CD007579. doi: 10.1002/14651858.CD007579.pub3. PMID 34002866
- [Derived] Kalava A, Darji SJ, Kalstein A, Yarmush JM, SchianodiCola J, Weinberg J. Efficacy of ginger on intraoperative and postoperative nausea and vomiting in elective cesarean section patients. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(2):184-8. doi: 10.1016/j.ejogrb.2013.02.014. Epub 2013 Mar 17. PMID 23510951

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment period: June 03, 2010 to April 12, 2011 Location: New York Methodist Hospital, Department of Obstetrics and Gynecology
Period: Overall Study
Arm/Group | Ginger | Placebo
Started | 116 | 123
Completed | 116 | 123
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ginger | Placebo | Total
Number analyzed (Participants) | 116 | 123 | 239
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 116 | 123 | 239
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.8 (5.3) | 33.0 (4.8) | 32.9 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 116 | 123 | 239
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 116 | 123 | 239

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Intra-operative and Post-operative Vomiting
Description: Participants who had intra-operative and post-operative vomiting were identified and compared between the two groups.
Time Frame: During surgery (1 hour) and thru 72 hours after surgery
Population: Number of participants who had vomiting in each group is compared to the other group using Chi square test
Measure: Count of Participants; unit: Participants
Arm/Group | Ginger | Placebo
Number analyzed (Participants) | 116 | 123
Participants | 30 | 45
Statistical Analysis 1: Comparison: Ginger vs Placebo; Number of participants who had vomiting in each group is compared to the other. Two sided Chi square test was conducted, Type I error of 0.05% and power of 80% are considered; Test type: Equivalence — Considering the null hypothesis that the number of participants who will have vomiting will be equal in the two arms, we performed this study with a significance level of 0.05% and power of 80% to prove that there is a difference in the number; p = 0.07, Chi-squared

ADVERSE EVENTS:
Groups:
- Placebo: 2 gm of placebo capsule
Arm/Group | Ginger | Placebo
All-Cause Mortality (participants affected / at risk) | 0/116 | 0/123
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/123
Other Adverse Events (participants affected / at risk) | 0/116 | 0/123

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes